CLINICAL TRIAL: NCT04478123
Title: An Open-Label, Pilot Study of Romiplostim for Conditioning Regimen-Related Thrombocytopenia After High-Dose Therapy and Autologous Hematopoietic Cell Transplantation
Brief Title: Using Romiplostim to Treat Low Platelet Counts Following Chemotherapy and Autologous Hematopoietic Cell Transplantation in People With Blood Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-180
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Results first posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2023-06

CONDITIONS: Multiple Myeloma; Hodgkin Lymphoma; Non-Hodgkin Lymphoma; HDT-AHCT
Keywords: High-Dose Therapy; Autologous Hematopoietic Cell Transplantation; Romiplostim; Thrombocytopenia; 20-180
MeSH Terms: conditions — Multiple Myeloma; Hodgkin Disease; Lymphoma, Non-Hodgkin; Thrombocytopenia | interventions — romiplostim

STUDY DESIGN:
Intervention Model Description: A single-center, open-label, pilot study of romiplostim for patients undergoing HDT-AHCT.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- romiplostim (Experimental): Patients will be enrolled prior to admission for High-Dose Therapy and Autologous Hematopoietic Cell Transplantation (HDT-AHCT), and they will undergo their planned HDT-AHCT for their respective hematologic malignancy as per institutional standards.
  Regardless of the conditioning regimen received, all patients will receive romiplostim 3.0 mcg/kg SC on Day +1 and romiplostim 2.0 mcg/kg SC on Day +8 after HDT-AHCT. Beyond Day +8, patients will be treated until platelet count is >50,000/mcL, without any platelet transfusions in the prior 48 hours. All doses after the second romiplostim dose will be titrated as per Table 3, based on weekly CBC/platelet counts. No patient will receive more than six doses of romiplostim, even if platelets have not corrected by Day +42.
  Interventions: Drug: Romiplostim

INTERVENTIONS:
Drug: Romiplostim — Romiplostim 3.0 mcg/kg SC on Day +1 and Romiplostim 2.0 mcg/kg SC on Day +8 after HDT-AHCT. Beyond Day +8, patients will be treated weekly until platelet count is >50,000/mcL, without any platelet transfusions in the prior 48 hours. All doses after the second Romiplostim dose will be titrated as per Table 3, based on weekly CBC/platelet counts. Patients will receive a maximum of six weekly doses of romiplostim.

SUMMARY:
The purpose of this study is to see if the study drug, romiplostim, helps low platelet count caused by the standard blood cancer treatment of chemotherapy and autologous hematopoietic cell transplantation. This study will also look at whether romiplostim can decrease the number of times the participant needs to return to the clinic for platelet transfusions to treat their low platelet count. In addition, the researchers will determine how safe it is to give romiplostim to people with blood cancer who have received treatment with chemotherapy and autologous hematopoietic cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years old diagnosed with multiple myeloma (MM), any subtype of Hodgkin lymphoma (HL), or any subtype of non-Hodgkin lymphoma (NHL)

  * For MM, the conditioning regimen used will be high-dose melphalan.°For HL and NHL, the conditioning will be one of the following high-dose regimens: BEAM, CBV, or TBC.
  * Other conditioning regimens not listed above, or variations of the above conditioning regimens, may be allowed at the discretion of the principal investigator if the regimen is considered myeloablative.
* Adequate organ function is required, defined as follows:

  * Serum bilirubin ≤ 2 mg/dL, unless benign congenital hyperbilirubinemia.
  * AST, ALT, and alkaline phosphatase < 3 times the upper limit of normal.
  * Creatinine clearance ≥ 40 ml/min (calculated by Cockcroft Gault)
  * LVEF ≥ 45% by MUGA or resting echocardiogram
  * Pulmonary function (FEV1 and corrected DLCO) ≥ 45% predicted.
  * Adequate performance status ECOG ≤ 2.
* Ability to provide written informed consent.
* Patients undergoing HDT-AHCT.

Exclusion Criteria:

* Patients with a previous diagnosis of a myeloid malignancy.
* Patients for whom the treating oncologist will be using a non-standard platelet transfusion threshold during the AHCT.
* Patients with a history of a prior symptomatic or incidental venous thromboembolic event (such as DVT or pulmonary embolism) within the prior 6 months are eligible if they are on and tolerating anti-coagulation, or greater than 6 months ago are eligible if they completed or are on and tolerating anti-coagulation.

  °A venous thrombotic event associated with a central venous catheter will not make the patient ineligible.
* Patients with a history of symptomatic arterial thrombotic events such as myocardial infarction, ischemic cerebral vascular accident or transient ischemic attack in the past 6 months are ineligible.
* Patients who had been diagnosed with Immune Thrombocytopenic Purpura (ITP) at any time prior to the AHCT are ineligible.
* Patients with a serious concomitant medical condition that could interfere with the conduct of the clinical trial, such as unstable angina, renal failure requiring hemodialysis, or active infection requiring IV antibiotics.
* Previous use of romiplostim, PEGylated recombinant human megakaryocyte growth and development factor, eltrombopag, recombinant human TPO, any other TPO receptor agonist, or any investigational platelet producing agent.
* Females who are pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 30 days after treatment discontinuation or longer if required by prescribing information for chemotherapy received during the study.
* Patients unwilling to use highly effective contraception during the study period and for the duration required by prescribing information for chemotherapy(ies) administered during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Scordo, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Scordo M, Gilbert LJ, Hanley DM, Flynn JR, Devlin SM, Nguyen LK, Ruiz JD, Shah GL, Sauter CS, Chung DJ, Landau HJ, Lahoud OB, Lin RJ, Dahi PB, Perales MA, Giralt SA, Soff GA. Open-label pilot study of romiplostim for thrombocytopenia after autologous hematopoietic cell transplantation. Blood Adv. 2023 Apr 25;7(8):1536-1544. doi: 10.1182/bloodadvances.2022007838. PMID 36409612
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Romiplostim: Patients will be enrolled prior to admission for High-Dose Therapy and Autologous Hematopoietic Cell Transplantation (HDT-AHCT), and they will undergo their planned HDT-AHCT for their respective hematologic malignancy as per institutional standards.
Period: Overall Study
Arm/Group | Romiplostim
Started | 62
Completed | 59
Not Completed | 3
Not completed — Pt withdrawal or refusal before begin prot txt | 2
Not completed — NE | 1

BASELINE CHARACTERISTICS:
Arm/Group | Romiplostim
Number analyzed (Participants) | 62
Age, Continuous [Median (Full Range); unit: years] | 63 [22 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 59
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 49
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 62

OUTCOME MEASURES:

1. Primary Outcome: Number of Days Post HDT-AHCT Requiring Transfusions or Grade 4 CTCAE Thrombocytopenia
Description: Common Terminology Criteria for Adverse Events (CTCAE) Version 5.
Time Frame: up to 42 days
Measure: Median (Full Range); unit: days
Arm/Group | Romiplostim
Number analyzed (Participants) | 59
days | 6 [0 to 17]

2. Secondary Outcome: Number of Platelet Transfusions Per Participant Issued During the AHCT Admission
Time Frame: up to 100 days from AHCT
Measure: Median (Full Range); unit: number of platelet transfusions per pt
Arm/Group | Romiplostim
Number analyzed (Participants) | 59
number of platelet transfusions per pt | 2 [0 to 7]

ADVERSE EVENTS:
Time Frame: Up to 42 days
Arm/Group | Romiplostim
All-Cause Mortality (participants affected / at risk) | 7/62
Serious Adverse Events (participants affected / at risk) | 0/62
Other Adverse Events (participants affected / at risk) | 62/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Romiplostim (N=62)
Lymphocyte count decreased (Investigations) | 62
Platelet count decreased (Investigations) | 62
White blood cell decreased (Investigations) | 62
Neutrophil count decreased (Investigations) | 53
Anemia (Blood and lymphatic system disorders) | 40
Blood bilirubin increased (Investigations) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/23/NCT04478123/Prot_SAP_000.pdf